CLINICAL TRIAL: NCT03761095
Title: A Phase 1B Study of Unesbulin (PTC596) in Combination With Dacarbazine in Patients With Locally Recurrent, Unresectable or Metastatic Relapsed/Refractory Leiomyosarcoma
Brief Title: A Study of Unesbulin (PTC596) in Combination With Dacarbazine in Participants With Advanced Leiomyosarcoma (LMS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC596-ONC-007-LMS
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma | interventions — PTC596; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Unesbulin and Dacarbazine (Experimental): Participants will receive unesbulin orally twice weekly in combination with dacarbazine IV once every 21 days. The first participant will receive dacarbazine 1000 mg/m^2 IV every 21 days in combination with unesbulin 200 mg tablet orally twice weekly. For subsequent participants, the dose level at which treatment is initiated will be selected based on the TITE-CRM using the most up to date dose DLT information from all participants previously treated. Participants will receive unesbulin 300 mg twice weekly in combination with dacarbazine in the expansion cohort. Treatment will continue for each participant until evidence of unacceptable toxicity, disease progression, or treatment discontinuation for another reason.
  Interventions: Drug: Unesbulin; Drug: Dacarbazine

INTERVENTIONS:
Drug: Unesbulin — Unesbulin will be administered as per the dose and schedule specified in the arm.
  Other Names: PTC596
Drug: Dacarbazine — Dacarbazine will be administered as per the dose and schedule specified in the arm.
  Other Names: DTIC

SUMMARY:
The primary objective of this study is to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of unesbulin in combination with dacarbazine for the treatment of advanced LMS and determine the overall safety profile of unesbulin in combination with dacarbazine.

This study will employ the time-to-event continual reassessment method (TITE-CRM) for dose finding. Treatment will be initiated at dose level 2 (DL2) (Dacarbazine 1000 milligrams per square meter [mg/m^2] intravenously [IV] every 21 days in combination with unesbulin 200 milligrams [mg] orally twice weekly) for the first participant. This dose level represents the investigator's best assessment of the MTD based on available toxicity data for both agents. For subsequent participants, the dose level at which treatment is initiated will be selected based on the TITE-CRM using the most up to date dose-limiting toxicity (DLT) information from all participants previously treated. To enroll additional participants at the RP2D, the study is amended to include an expansion cohort of up to 12 participants (some of whom could be ongoing participants who reconsent).

Treatment will continue for each participant until evidence of unacceptable toxicity, disease progression, or treatment discontinuation for another reason.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent of an Institutional Review Board (IRB)-approved informed consent form (ICF) and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information (if appropriate).
2. Willingness and ability to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.
3. Disease Status including all of the following:

   1. Histological or cytological confirmation of LMS arising at any anatomic site.
   2. Advanced (metastatic) or locally advanced unresectable disease.
   3. Ineligible for other high-priority national or institutional study.
   4. Measurable disease per RECIST v1.1 criteria.

   Demographics:
4. Age greater than or equal to (>/=) 18
5. Male and Female

   Performance Status:
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.

   Hematopoietic:
7. Absolute neutrophil count (ANC) count >/= 1,500/cubic millimeters (mm^3) without the use of growth factors in the past 7 days;
8. Platelet count >=100,000/mm^3 without platelet transfusion in the past 5 days;
9. Hemoglobin >=9 grams per deciliter (g/dL) (packed red blood cell transfusion is allowed).

   Hepatic:
10. Bilirubin lesser than (<) upper limit of normal (ULN);
11. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <1.5 times ULN;
12. Participants with liver metastases may be enrolled.

    Pulmonary:
13. Participants with well-controlled asthma (for example Use of rescue medications <2 times/week over the last 12 months) or Chronis Obstructive Pulmonary Disease (COPD) (for example no exacerbations over the prior 3 months) may be enrolled.

    Renal:
14. Creatinine <1.5 times normal, or creatinine clearance greater than (>) 45 milliliters per minute (mL/min).

    Prior Therapies:
15. Toxicity from prior therapies recovered to Grade lesser than or equal to (<=) 1 or participant's baseline, except for alopecia. In addition, endocrinopathies associated with prior immunotherapy based treatments which are well controlled on replacement medication are not exclusionary
16. Chemotherapy:

    a. Up to and inclusive of 4 prior systemic cytotoxic oncology therapy regimens for metastatic, locally recurrent, or unresectable LMS, with the last dose of prior therapy administered no fewer than 30 days or 5 times the drug half-life prior to screening. Note: prior treatment with non-cytotoxic therapy regimens (for example targeted therapies, hormonal therapies, or tyrosine kinase inhibitors) are not considered cytotoxic oncology therapies.

    Surgery:
17. At least 4 weeks since prior surgery and recovered in opinion of investigator.

    Other:
18. Capable of swallowing oral medication.
19. Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy.
20. Males and females of childbearing potential must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 90 days after treatment discontinuation. Note: The Definition of effective contraception will be based on the judgement of the Principal Investigator (PI) or Designee.

Exclusion Criteria:

Participants meeting any of the following criteria will not be eligible for enrollment:

1. Received any systemic anticancer therapy including investigational agents <=3 weeks prior to initiation of study treatment. Additionally, Participants may have not received radiation </= 3 weeks prior to initiation of study treatment.
2. Co-existing active infection or any co-existing medical condition likely to interfere with study procedures, including:

   a. Significant cardiovascular disease (New York Heart Association Class III or IV cardiac disease), myocardial infarction within the past 6 months, unstable angina, congestive heart failure requiring therapy, unstable arrhythmia or a need for anti-arrhythmic therapy, or evidence of ischemia on electrocardiogram (ECG), marked baseline prolongation of QT/QTc (corrected QT interval) interval, for example, repeated demonstration of a QTc interval >500 milliseconds (msec) (Long QT Syndrome [congenital]).
3. Known human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) positivity.
4. History of solid organ transplantation.

   Therapeutics:
5. Known or suspected allergy or immediate or delayed hypersensitivity to unesbulin or dacarbazine or any agent given in this study.

   Gastrointestinal:
6. Bowel obstruction, malabsorption, or other contraindication to oral medication.
7. Gastrointestinal disease or other condition that could affect absorption.
8. Active peptic ulcer disease.
9. Inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis.
10. Any condition that impairs participant's ability to swallow oral medications.

    Wounds /Surgery:
11. Serious non-healing wound, ulcer, or bone fractures.
12. Major surgery, open biopsy or significant traumatic injury which has not recovered in the opinion of the investigator, within 28 days of baseline.
13. Mucosal or internal bleeding.

    Concomitant Medications:
14. Concomitant strong CYP1A2 inhibitors (like selective serotonin reuptake inhibitor [SSRI] agents fluvoxamine and fluoxetine) should be avoided. CYP1A2 inhibitors may inhibit the conversion of dacarbazine to its active metabolite and may increase the exposure of unesbulin.

    Other:
15. Prior malignancies other than LMS, that required treatment or have shown evidence of recurrence (except for non-melanoma skin cancer or adequately treated cervical carcinoma in situ) during the 5 years prior to initiation. Cancer treated with curative intent more than 5 years previously and without evidence of recurrence is not an exclusion.
16. Known coagulopathy or bleeding diathesis. Participants on anti-coagulation should be monitored closely and International Normalized Ratio (INR) within normal range.
17. Prior or ongoing clinically significant illness, medical or psychiatric condition, medical history, physical findings, ECG findings, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the participant, or alter the absorption, distribution, metabolism, or excretion of the study drugs, or could impair the assessment of study results.
18. History of brain metastases or leptomeningeal disease at any time in participant's history, including treated central nervous system (CNS) disease which is clinically and radiographically stable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
MTD and RP2D of Unesbulin in Combination With Dacarbazine | First 2 cycles of treatment (6 weeks)
  MTD will be determined using the TITE-CRM for dose-finding. MTD is defined as the dose associated with a target probability of DLT of 0.25.
Number of Participants With Adverse Events | From screening until end of study (up to approximately 1.5 years)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (Percentage of Participants With Objective Response) as Determined by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | From Baseline until the date of objectively documented progression per RECIST v1.1 or the date of initiation of subsequent therapy or palliative local therapy, whichever occurs first (up to approximately 1.5 years)
  Objective Response is defined as confirmed best response of complete response (CR) or partial response (PR).
Time to Response as Determined by the Investigator Using RECIST v1.1 | From Baseline until the date of first occurrence of CR or PR (up to approximately 1.5 years)
  Time to response is defined as the first time either PR or CR occurs.
Duration of Response (DOR) | Time from the date of first confirmed response to the date of the first documented tumor progression or death due to any cause, whichever occurs first (up to approximately 1.5 years)
  DOR is defined as the time from the date of first confirmed response to the date of the first documented tumor progression (per RECIST v1.1) or death due to any cause, whichever occurs first.
Progression-Free Survival (PFS) | Time from the first dose of study drug to the date of the first documented tumor progression or death due to any cause, whichever occurs first (up to approximately 1.5 years)
  PFS is defined as the time from the first dose of study drug to the date of the first documented tumor progression as determined by the investigator using RECIST v1.1 or death due to any cause, whichever occurs first.
Best Overall Response Rate (Disease Control Rate) (Percentage of Participants With Best Overall Response) | From Baseline until the date of objectively documented progression per RECIST v1.1 or the date of initiation of subsequent therapy or palliative local therapy, whichever occurs first (up to approximately 1.5 years)
  Best overall response is defined as CR, PR and stable disease (SD).
Overall Survival (OS) | Time from the first dose of study drug to the date of death from any cause (up to approximately 1.5 years)
  OS is defined as the time from the first dose of study drug to the date of death from any cause.
Maximum Observed Plasma Concentration (Cmax) of Unesbulin, Dacarbazine, and Inactive Metabolite of Dacarbazine (5-amino-imidazole-4-carboxamide [AIC]) | Unesbulin: Predose (within 1 hour [hr]); 1,2,3 to 824, 48, 72 hrs postdose (during any cycle); Dacarbazine and AIC: Predose (within 1 hr); 0.5,1 hr post start of infusion; 0.25,0.5,1,3,7,23 hrs postdose on Cycle 1 Day 1,Cycle 2 Day 1 (each cycle=21 days)
  Pharmacokinetic (PK) variables will be calculated from the plasma concentration data using standard compartmental or non-compartmental methods, as appropriate for the data.
Time to Reach Maximum Plasma Concentration (Tmax) of Unesbulin, Dacarbazine, and Inactive Metabolite of Dacarbazine (AIC) | Unesbulin: Predose (within 1 hr); 1,2,3 to 824, 48, 72 hrs postdose (during any cycle); Dacarbazine and AIC: Predose (within 1 hr); 0.5,1 hr post start of infusion; 0.25,0.5,1,3,7,23 hrs postdose on Cycle 1 Day 1,Cycle 2 Day 1 (each cycle=21 days)
  PK variables will be calculated from the plasma concentration data using standard compartmental or non-compartmental methods, as appropriate for the data.
Area Under the Plasma Concentration-Time Curve (AUC) of Unesbulin, Dacarbazine, and Inactive Metabolite of Dacarbazine (AIC) | Unesbulin: Predose (within 1 hr); 1,2,3 to 824, 48, 72 hrs postdose (during any cycle); Dacarbazine and AIC: Predose (within 1 hr); 0.5,1 hr post start of infusion; 0.25,0.5,1,3,7,23 hrs postdose on Cycle 1 Day 1, Cycle 2 Day 1 (each cycle=21 days)
  PK variables will be calculated from the plasma concentration data using standard compartmental or non-compartmental methods, as appropriate for the data.
Half-Life (t1/2) of Unesbulin, Dacarbazine, and Inactive Metabolite of Dacarbazine (AIC) | Unesbulin: Predose (within 1 hr); 1,2,3 to 824, 48, 72 hrs postdose (during any cycle); Dacarbazine and AIC: Predose (within 1 hr); 0.5,1 hr post start of infusion; 0.25,0.5,1,3,7,23 hrs postdose on Cycle 1 Day 1, Cycle 2 Day 1 (each cycle=21 days)
  PK variables will be calculated from the plasma concentration data using standard compartmental or non-compartmental methods, as appropriate for the data.
Apparent Clearance (CL/F) of Unesbulin, Dacarbazine, and Inactive Metabolite of Dacarbazine (AIC) | Unesbulin: Predose (within 1 hr); 1,2,3 to 824, 48, 72 hrs postdose (during any cycle); Dacarbazine and AIC: Predose (within 1 hr); 0.5,1 hr post start of infusion; 0.25,0.5,1,3,7,23 hrs postdose on Cycle 1 Day 1, Cycle 2 Day 1 (each cycle=21 days)
  PK variables will be calculated from the plasma concentration data using standard compartmental or non-compartmental methods, as appropriate for the data.
Apparent Volume of Distribution (Vz/F) of Unesbulin, Dacarbazine, and Inactive Metabolite of Dacarbazine (AIC) | Unesbulin: Predose (within 1 hr); 1,2,3 to 824, 48, 72 hrs postdose (during any cycle); Dacarbazine and AIC: Predose (within 1 hr); 0.5,1 hr post start of infusion; 0.25,0.5,1,3,7,23 hrs postdose on Cycle 1 Day 1, Cycle 2 Day 1 (each cycle=21 days)
  PK variables will be calculated from the plasma concentration data using standard compartmental or non-compartmental methods, as appropriate for the data.
Accumulation Ratio (R) of Unesbulin, Dacarbazine, and Inactive Metabolite of Dacarbazine (AIC) | Unesbulin: Predose (within 1 hr); 1,2,3 to 824, 48, 72 hrs postdose (during any cycle); Dacarbazine and AIC: Predose (within 1 hr); 0.5,1 hr post start of infusion; 0.25,0.5,1,3,7,23 hrs postdose on Cycle 1 Day 1, Cycle 2 Day 1 (each cycle=21 days)
  PK variables will be calculated from the plasma concentration data using standard compartmental or non-compartmental methods, as appropriate for the data.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Mayo Clinic Florida, Jacksonville, Florida
  - John Hopkins, Baltimore, Maryland
  - Washington University Medical Campus, St Louis, Missouri
  - Columbia University Medical Center, New York, New York

REFERENCES:
- [Derived] Van Tine BA, Ingham MA, Attia S, Meyer CF, Baird JD, Brooks-Asplund E, D'Silva D, Kong R, Mwatha A, O'Keefe K, Weetall M, Spiegel R, Schwartz GK. Phase Ib Study of Unesbulin (PTC596) Plus Dacarbazine for the Treatment of Locally Recurrent, Unresectable or Metastatic, Relapsed or Refractory Leiomyosarcoma. J Clin Oncol. 2024 Jul 10;42(20):2404-2414. doi: 10.1200/JCO.23.01684. Epub 2024 Apr 29. PMID 38684039
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217411&parentIdentifier=PTC596-ONC-007-LMS&attachmentIdentifier=d3fd6143-2549-49e7-a4e6-bc948b6ca931&fileName=PTC596-ONC-007-LMS_Protocol_Update_Offline_approval_by_Mark.pdf&versionIdentifier=